CLINICAL TRIAL: NCT01732991
Title: Assessing the Impact of the Prostatic Photo-vaporization (PVP) With Greenlight Laser Using Prostatic MRI and Contrast-enhanced Ultrasound
Brief Title: Assessing the Impact of the PVP With Greenlight Laser Using Prostatic MRI and Contrast-enhanced Ultrasound
Acronym: PROPIL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Tours (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PHAO 2012 - FB / PROPIL
Record Dates: First submitted 2012-11-19; First posted 2012-11-26 (Estimated); Last update posted 2025-12-26 (Actual); Status verified 2015-08

CONDITIONS: Prostatic Hypertrophy, Benign
Keywords: Prostatic Hypertrophy, Benign; Greenlight laser; Prostatic photovaporization; Prostatic MRI; Prostatic contrast-enhanced ultrasound; Urinary irritative signs; Postoperative necrotic area
MeSH Terms: conditions — Prostatic Hyperplasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- prostatic photo-vaporization (Experimental): prostatic photo-vaporization (PVP) surgery with laser Greenlight
  Interventions: Device: prostatic photo-vaporization (PVP)

INTERVENTIONS:
Device: prostatic photo-vaporization (PVP) — Prostatic photo-vaporization using a lithium laser of 532nm wavelength (GREEN-LIGHT XPS™,American Medical Systems, Minnetonka, MN, USA) emitting by a fiber MoXy™ a maximum power of 180 W continuously. Using common practice and according to the CE labelling.

SUMMARY:
The PVP by Greenlight laser 180W is becoming a potential therapeutic alternative in the treatment of benign prostatic hypertrophy (BPH) as recommended.

The PVP creates a prostatic box after the vaporization of the prostatic tissue of BPH. The underlying prostatic tissue is the site of an ischemic necrosis secondary to the thermal effects of proximity of the PVP. We intend to measure by prostatic MRI and contrast-enhanced ultrasound the necrosis.

DETAILED DESCRIPTION:
The laser PVP with an optical fiber firing side carries out a vaporization of next prostatic tissue and a necrosis of underlying prostatic tissue which corresponds to a postoperative inflammatory area.

One of the side effects of this technique is the irritative syndrome which may involve urinary frequency, urgency or burning urination in approximately 10 to 20% at 1 month.

The current literature does report neither the analysis of the underlying inflammatory necrotic area in prostatic vaporized tissue, nor the analysis of the urinary irritative signs post-laser PVP.

Progresses in the field of functional ultrasound imaging allow us to consider a study of evolution of the underlying necrotic area devoid of micro-vascularisation under effect of PVP laser. The parallel with results of MRI (radiological technique most referenced) during the same period would help to support the experimental results of prostatic contrast-enhanced ultrasound.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 40 years old without an upper age limit
* Informed orally and in writing, having signed a consent which match to the research
* Patient with a benign prostatic hypertrophy requiring surgical treatment by PVP
* Person affiliated to a social security system

Exclusion Criteria:

* Contraindications to MRI for patients with:

  * ocular metallic foreign object
  * any electronic medical device implanted by irremovable way (pacemakers, neuro-stimulator, cochlear implants ...)
  * metallic heart valve, old heart valves are specially an absolute contraindication because of risk of dysfunction
  * vascular clips implanted formerly on brain aneurysm
* Allergy to Gadolinium
* Contraindications to the contrast medium Sonovue:

  * Hypersensitivity to hexafluorinated sulphur or any other components of Sonovue
  * Recent acute coronary syndrome (within 6 months before the intervention)
  * Unstable ischemic heart disease (myocardial infarction being formed or evolving, typical angina of rest in the previous month)
  * Significant worsening of cardiac symptoms between the pre anaesthesia consultation and intervention
  * Recent intervention (less than 6 months) on coronary arteries or other factor suggesting clinical instability (changes in ECG, changes in clinical or biological parameters)
  * Acute heart failure or heart failure stage III or IV
  * Severe arrhythmias
  * Right-left shunt
  * Acute endocarditis
  * Valve prothesis
  * Severe pulmonary hypertension (pulmonary artery pressure > 90mmHg)
  * Systemic hypertension uncontrolled
  * Respiratory distress syndrome
* Prostatic biopsy < 30 days or anal pathology
* Patient with prostate cancer
* Patient with a urinary infection
* Patient with preoperative urinary catheter
* Patient with a contraindication for surgery
* Adult patient with a legal protection measure

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2012-09; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Evolution of thickness of the average necrotic area | J0 (immediately after surgery) M1, M6 and M12
  The primary outcome measure is the measurement of the thickness of the average necrotic area in millimeters on prostatic monitoring MRI and contrast-enhanced ultrasound (no hypothesis in this descriptive study). The variables will be collected immediately after surgery as well as M1, M6 and M12.

SECONDARY OUTCOMES:
Evolution of urinary irritative signs over 12 months | J0, M1, M6 and M12
  Evolution of urinary irritative signs over 12 months (prostatic monitoring MRI and contrast-enhanced ultrasound): score of IPSS questionary, results of the examination (binary variable)
Evolution of prostatic volume over 12 months | J0, M1, M6 and M12
  Evolution of prostatic volume over 12 months (prostatic monitoring MRI and contrast-enhanced ultrasound)

CONTACTS AND LOCATIONS:
Overall Officials: Franck BRUYERE, MD, Principal Investigator — CHRU TOURS
Locations (1):
- Chru Tours, Tours, France

REFERENCES:
- [Result] Bruyere F, Bodin T, Bleuzen A, Patat F, Brunereau L. Penetration depth with the XPS GreenLight laser assessed by contrast enhanced ultrasonography. J Endourol. 2013 Oct;27(10):1282-6. doi: 10.1089/end.2013.0368. Epub 2013 Aug 21. PMID 23837622